CLINICAL TRIAL: NCT02406924
Title: Maxillary Horizontal and Vertical Bone Augmentation Using Particulated Biomaterial Associated With Autogenous Bone, Covered and Stabilized by a Collagen Membrane and Pins
Brief Title: Bone Augmentation Using Particulated Biomaterial and Autogenous Bone, Stabilized by Collagen Membrane and Pins (PaMP)
Acronym: PaMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pedro Tortamano (Other)
Responsible Party: Sponsor-Investigator, Pedro Tortamano, PHD, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UniversidadeSP
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-04

CONDITIONS: Alveolar Bone Grafting; Bone Augmentation
Keywords: pin; particulated graft; bone augmentation; vertical augmentation; horizontal augmentation
MeSH Terms: conditions — Prostatic Intraepithelial Neoplasia | interventions — Biopsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sausage graft (Experimental): Bone graft performed with a mixture of particulated autogenous and lyophilized bovine bone, stabilized with collagen membrane and pins.
  Interventions: Procedure: Biopsy; Radiation: Computerized Tomography; Other: Standardized periapical radiographs; Other: Intraoral scanning
- Bone block graft (Active Comparator): Bone graft performed with a block of autogenous bone stabilized by a screw associated with lyophilized bovine bone and collagen membrane.
  Interventions: Procedure: Biopsy; Radiation: Computerized Tomography

INTERVENTIONS:
Procedure: Biopsy — A cylinder of grafted bone will be removed from the location elected for the implant installation with an appropriate trephine
Radiation: Computerized Tomography — An initial computerized tomography will be made before the first surgery, and a final computerized tomography will be made after 9 months, previously to the second surgery
Other: Standardized periapical radiographs — A device will be adopted for the standardization, and radiographs will be taken at day 0, 3 months, 6 months, 12 months, 18 months, 24 months after implant installation
  Arms: Sausage graft
Other: Intraoral scanning — Intraoral scanning will be made before the graft, at implant installation, 3 months, 6 months, 12 months, 18 months, 24 months after implant installation
  Arms: Sausage graft

SUMMARY:
Twenty four patients with bone resorption on the anterior maxilla will be divided into two groups with different kinds of grafting: bone block associated with particulated biomaterial and particulated mixture of autogenous bone and biomaterial stabilized by collagen membrane and pins. The techniques will be compared according to volume gain, quality of graft osseointegration, implant survival and maintenance of the level of soft tissues.

DETAILED DESCRIPTION:
Twenty four patients will be selected analysing the resorption on the front maxilla and will be divided into two groups. Experimental group will receive a particulated mixture of autogenous and lyophilized bovine bone, stabilized with a collagen membrane and pins over the vertical and/or horizontal defect, while Control group will receive a bone block graft, stabilized with fixation screws , covered with lyophilized bone and a collagen membrane. After a period of nine months, the volume increase will be measured trough the difference found between the initial computerized tomography and the final computerized tomography.

Dental implants will be placed according to the prosthetic need and bone cylinders will be removed from the respective location. The cylinders will be histologically analysed in order to verify the quality of the graft osteointegration. After the prosthesis installation, the implant survival and the soft and hard tissues will be followed up for a minimum period of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* absence of teeth at anterior maxilla
* need of vertical or horizontal bone reconstruction at anterior maxilla

Exclusion Criteria:

* smoking habits
* diabetes
* systemic diseases which interfere with osseous metabolism
* active periodontal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-12 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
vertical gain | 9 months
  Measures will be taken from computerized tomography in axial sections
horizontal gain | 9 months
  Measures will be taken from computerized tomography in transverse sections
implants survival | 24 months
  Clinical examination and standardized radiographs will be taken periodically
soft tissue volume | 24 months
  Measures will be taken from images generated by intraoral scanning in an occlusal view

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Tortamano, PHD, Principal Investigator — University of Sao Paulo